CLINICAL TRIAL: NCT01664715
Title: A Randomized Trial of Recommendations for Exercise to Prevent Weight Regain
Acronym: POWeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSCL19775; R01HL111842 (NIH)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Overweight; Obesity; Weight Loss
Keywords: Overweight; Obesity; Exercise; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 150 Minutes per Week (Active Comparator): Performs 150 minutes of physical activity per week.
  Interventions: Behavioral: 150 Min/Week
- 225 Minutes per Week (Active Comparator): Performs 225 minutes of physical activity per week.
  Interventions: Behavioral: 225 Min/Week
- 300 Minutes per Week (Active Comparator): Performs 300 minutes of physical activity per week.
  Interventions: Behavioral: 300 Min/Week

INTERVENTIONS:
Behavioral: 150 Min/Week — Performs 150 min/wk of planned moderate intensity aerobic exercise.
  Arms: 150 Minutes per Week
Behavioral: 225 Min/Week — Performs 225 min/wk of planned moderate intensity aerobic exercise.
  Arms: 225 Minutes per Week
Behavioral: 300 Min/Week — Performs 300 min/wk of planned moderate intensity aerobic exercise.
  Arms: 300 Minutes per Week

SUMMARY:
The investigators will conduct a randomized trial to evaluate the effectiveness of 3 levels of recommended exercise in initially overweight and obese sedentary men and women on the prevention of weight regain. Participants will complete a 3 mo. weight loss intervention of decreased energy intake (EI) and increased energy expenditure (100 minutes of physical activity per week). Participants achieving clinically significant weight loss (> 5% of initial weight), will be randomly assigned to 12 mos. of exercise at levels of energy expenditure of exercise (EEEx) recommended by Health and Human Services (HHS), American College of Sports Medicine(ACSM), Institute of Medicine (IOM): 150, 225, or 300 minutes per week. Major outcome assessments will occur prior to weight loss (-3 mos.), at completion of weight loss (0 mos.), at the midpoint (6 mos.), and completion of weight maintenance (12 mos.).

DETAILED DESCRIPTION:
The investigators propose a randomized trial in 287 overweight and obese, sedentary adults (at least 50% women). Participants achieving clinically significant weight loss (≥5%) following a 3 mo. reduced energy diet and a program of PA (100 min/wk) will be randomly assigned to either maintain exercise at 150 min/wk. or increase exercise to 225 min/wk or 300 min/wk. while consuming a weight gain prevention diet over a 12 mo. period. Exercise will be verified (combination of on-site and HR monitor) and EEEx will be measured at 5 mo. intervals beginning at mo. 5. In-person behaviorally based clinic meetings will be conducted weekly during the 3 mo. weight loss period (-3 to 0 mos.) and during the first 3 mos. of the weight regain prevention period. During the final 9 mos. of weight regain prevention, clinics will be held bi-monthly using group conference calls. We have not proposed to randomize participants to a true control group (i.e. no exercise or diet) following the 3 mo. weight loss program as published data indicates significant weight regain in individuals receiving no follow-up treatment after weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 55 years.
* BMI of 25 to 45.0.
* Clearance for participation from their Primary Care Physician (PCP)

Exclusion Criteria:

* Participation in a research project involving weight loss or exercise in the previous 6 mos., as these proximal experiences may impact the results of this study.
* Participation in a regular exercise program (i.e., > 500 kcal/wk. of planned activity as estimated by questionnaire)
* Not weight stable (+ or - 4.5 kg) for 3 mos. prior to intake.
* Unwilling to be randomized to 1 of 3 exercise groups subsequent to weight loss.
* Pregnant during the previous 6 mos., lactating, or planned pregnancy in the following 15 mos.
* Serious medical risk such as type 1 diabetes, cancer, recent cardiac event (i.e., heart attack, angioplasty, etc.). This is determined by the individual's physician via the clearance to participate in the investigation and the health history (Appendix) interpreted by the staff physician.
* Eating disorders as determined by the Eating Attitudes Test using a score of 20 or greater
* Current treatment for psychological problems, or taking psychotropic medications
* Medications known to significantly affect weight (gain or loss).
* Adherence to specialized diet regimens, i.e., multiple food allergies, vegetarian, macrobiotic, etc.
* Do not have access to grocery shopping and meal preparation (i.e. those in military, college with cafeteria plan, etc.).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 287 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Prevention of Weight Regain | 12 Months
  To compare the effectiveness of 3 exercise recommendations on the prevention of weight regain over 12 mos. subsequent to clinically significant weight loss (> 5%). We expect participants will regain weight in a dose-response manner, i.e. greatest, intermediate and least weight regain for the 150, 225, and 300 minute. groups, respectively.
Gender Differences in Weight Regain | 12 Months
  To evaluate gender differences in weight regain over 12 months in response to 3 exercise recommendations. Based on available preliminary data we expect men will regain less weight than women.

SECONDARY OUTCOMES:
Compensatory Changes to three exercise levels | 12 Months
  Evaluating the impact of potential compensatory changes in daily physical activity and energy intake on weight regain in response to 3 exercise recommendations. Any observed compensatory responses would inform the development of subsequent targeted interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, EdD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas - Robinson Hall, Lawrence, Kansas, United States

REFERENCES:
- [Derived] Kracht CL, Brown DMY, Gorczyca AM, Jakicic JM, Szabo-Reed A, Washburn R, Donnelly JE. Association Between Wake-Time Movement Behaviors and Weight Loss Maintenance. Obesity (Silver Spring). 2025 Nov 16:10.1002/oby.70082. doi: 10.1002/oby.70082. Online ahead of print. PMID 41243427
- [Derived] Szabo-Reed AN, Martin LE, Savage CR, Washburn RA, Donnelly JE. Pre-post intervention exploring cognitive function and relationships with weight loss, intervention adherence and dropout. Health Psychol Behav Med. 2023 Jan 6;11(1):2162528. doi: 10.1080/21642850.2022.2162528. eCollection 2023. PMID 36632603
- [Derived] Szabo AN, Washburn RA, Sullivan DK, Honas JJ, Mayo MS, Goetz J, Lee J, Donnelly JE. The Midwest Exercise Trial for the Prevention of Weight Regain: MET POWeR. Contemp Clin Trials. 2013 Nov;36(2):470-8. doi: 10.1016/j.cct.2013.08.011. Epub 2013 Sep 4. PMID 24012915